CLINICAL TRIAL: NCT05393947
Title: Investigation of the Effect of the Training Given According to Orem's Self-Care Deficit Theory Based Education on the Management of Chemotherapy Side Effects and Improving the Patient's Self-Care of the Patients With Breast Cancer
Brief Title: Investigation of the Effect of Education on Symptom Management on Symptom Management in Patients With Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Dilek Urtekin, Principal Investigator, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SaglikBilimleriU_DU
Record Dates: First submitted 2022-05-18; First posted 2022-05-26 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Patient Education as Topic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient aducation (Experimental): It is planned to provide education to patients about the side effects of chemotherapy.
  Interventions: Other: patient education
- observation (No Intervention): While training the patients in the intervention group, observations will be made on the patients in the experimental group.

INTERVENTIONS:
Other: patient education — It is planned to provide education to patients about the side effects of chemotherapy.
  Arms: patient aducation

SUMMARY:
It is used with different treatment options such as chemotherapy, radiotherapy and surgery in the treatment of breast cancer, which is common in women among all cancers in the world. Side effects such as nausea, vomiting, neuropathy, oral nucositis, constipation, sleep problems, fatigue and alopecia occur due to chemotherapeutic agents applied in the treatment of breast cancer. Due to the lack of information and side effects related to cancer treatment, it negatively affects the adherence to treatment and self-care power of individuals. In this study, it was planned to examine the effect of training given for chemotherapy-related symptoms on self-care power and the management of chemotherapy side effects. Your study was planned as a single-center, randomized controlled quasi-experimental design. The research sample will consist of breast cancer patients aged between 18 and 65 years who were treated at Tekirdağ Namık Kemal University Hospital between July 2022 and April 2023 and accepted to participate in the study [26 intervention (experimental) group - 26 control group]. Intervention and control groups will be determined by using the random numbers table from the simple random sampling method, which is one of the probability sampling methods. In line with Orem's Self-Care Deficit Theory, a training booklet will be created for the management of chemotherapy side effects. Participants in the intervention (experimental) group of the study will be given training on chemotherapy side effects, which lasts 20-30 minutes at the first interview. Patient Information Form, Nightingale Symptom Evaluation Scale and Self-Care Behaviors Inquiry Form will be filled. Patients will be followed up for a total of 5 times during 4 cycles of chemotherapy and will be interviewed face-to-face at each chemotherapy cycle. Data collection tools will be filled in face-to-face interviews, the patient's side effects due to chemotherapy and the methods applied in the face of these side effects will be questioned, suggestions will be given for the control of chemotherapy side effects, and the patient's questions will be answered. No intervention will be applied to the participants in the control group of the study. In this study, it is thought that education and follow-up based on Orem's Self-Care Deficit Theory will contribute to the development of self-care behaviors and effective side-effect management in patients receiving chemotherapy for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Receiving adjuvant chemotherapy with the diagnosis of breast cancer,
* Receiving CE (cyclophosphamide-epirubicin) or CA (cyclophosphamide-adriamycin) treatment protocol,
* First time receiving chemotherapy,
* Aged between ≥ 18 and ≤ 65,
* Can understand Turkish and can read and write,
* Those whose health status is suitable for participating in the research,
* Having stage I, stage II and stage III breast cancer,
* Identified as patients who volunteered to participate in the study

Exclusion Criteria:

* Metastasis detected
* Those with a diagnosis of psychiatric disease
* Those who want to leave the research and
* Patients whose general condition deteriorates will not be included in the study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Symptom management | 3 weeks
  A training booklet on the management of chemotherapy side effects was prepared for the intervention (experimental) group of the study, based on Orem's Self-Care Disability Theory. Before the first chemotherapy course, a training was given in parallel with the training booklet. The training booklet was given to the patients. This training and education booklet contributed to the management of chemotherapy-related side effects and the development of self-care behaviors in individuals with breast cancer at the end of 4 chemotherapy cycles.

SECONDARY OUTCOMES:
Nightingale Symptom Assessment Scale | 3 weeks
  The Nightingale Symptom Assessment Scale is a quality of life scale developed for cancer patients. It measures the level of being affected by the disease/treatment-related problems of the patients. This scale was scored as "0" if the patient's response to the item being evaluated was no, and "4" if it was too much. O point stated that the quality of life was not affected at all, and 4 points stated that it was greatly affected.
Self-Care Behaviors Inquiry Form | 3 weeks
  The Self-Care Behaviors Inquiry Form was prepared by the researchers in order to question the individual's self-care behaviors. The form consists of questions about the patient's daily life self-care behaviors related to chemotherapy-induced nausea-vomiting, changes in taste and smell, oral mucositis, diarrhea, constipation, fatigue, sleep problems and alopecia. This form was applied in the form of individuals answering the statements themselves. Response options were answered with 0 points for the answer "I never apply" and 3 points for the answer "I always apply". High scores showed that the patient's self-care behaviors improved positively.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek URTEKİN, Principal Investigator — İstanbul Health Sciences University
Locations (1):
- Saglik Bilimleri Universitesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No